## **OFFICIAL TITLE:**

THE EFFECTS OF PROBIOTICS ON METABOLIC BIOMARKERS, INFLAMMATION, AND THE ANTIOXIDANT SYSTEM IN PATIENTS WITH TYPE 2 DIABETES MELLITUS

Date: 17.04.2018

## **Statistical Analysis Plan (SAP)**

Statistical analysis was performed using SPSS 25.0 statistical package program. Data from all patients who completed the study were included in the statistical analysis. For descriptive findings, categorical variables were presented as numbers and percentages, and continuous variables were presented as mean, standard deviation, minimum value and maximum value. Kolmogorov-Smirnov normality tests were used to determine whether the data showed normal distribution. Pearson chi-square test was used to analyse categorical variables. Parametric tests (t test in independent groups, t test in dependent groups) were used in the analysis of normally distributed data, and non-parametric tests (Mann-Whitney U test, Wilcoxon Signed Rank Test) were used in the analysis of non-normally distributed data. Statistical significance level was accepted as p<0.05.